CLINICAL TRIAL: NCT05266235
Title: Clinical Validation of the Withings ECG Monitor for the Detection of Atrial Fibrillation
Acronym: QDA-UE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02730-41
Record Dates: First submitted 2022-02-09; First posted 2022-03-04 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Withings WBS08 and 12-lead reference ECG (Experimental): The electrodes of the 12-lead ECG will be set up on the participants, before they step on withings WBS08 to have ECGs simultaneously recorded by the study device and the control device
  Interventions: Device: Validation of the Withings bodyscan scale WBS08

INTERVENTIONS:
Device: Validation of the Withings bodyscan scale WBS08 — Participants will undergo simultaneous recordings of ECGs with the comparator and the study device

SUMMARY:
The aim of the study is to demonstrate the performance of Withings WBS08 in the automatic identification of atrial fibrillation and sinus rhythm.

DETAILED DESCRIPTION:
Patients included will be those presenting for consultation in the various participating clinical services. For each patient, an ECG will be recorded with the WBS08 and with the reference device Cardiovit FT1, at rest and after an exercise session.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 18 years of age or older
* Subject able to read, understand and provide written informed consent
* Subject willing and able to participate in the study procedures as described in the consent form
* Subject able to communicate effectively with and willing to follow instructions from the study staff
* Subject affiliated to a social security system

For subjects enrolled into the AF population, subjects must have a known diagnosis of AF and be in AF at the time of screening. Subjects may have any type of AF including paroxysmal, persistent, and permanent AF.

Exclusion Criteria:

* Vulnerable subject with regard to regulations in force :
* Subject who is deprived of liberty by judicial, medical or administrative decision,
* Underage subject,
* Legally protected subject, or subject who is unable, linguistic or psychic incapacity, to sign the written informed consent form
* Subject within several of the above categories
* Subject who refused to participate in the study
* Subject mentally impaired resulting in limited ability to cooperate
* Subject with a pacemaker, ICD (Implantable cardioverter defibrillator) or other implanted electronic stimulator
* Patient with pathologic disorder that may affect motricity resulting in significant tremor that prevents subject from being ablle to hold still (e.g Parkinson disease)
* Patient unable to stay in an upright position for the duration of study measures
* Acute myocardial infarction (MI) within 90 days of screening or other cardiovascular disease that, in the opinion of the investigator, may increase the risk to the subject or renders data uninterpretable (e.g. recent or ongoing unstable angina, decompensated heart failure, active myocarditis or pericarditis)
* Acute pulmonary embolism or pulmonary infarction, within 90 days of screening
* Stroke or transient ischemic attack within 90 days of screening
* Active life-threatening rhythms as determined by the investigator (ventricular tachycardia, ventricular fibrillation, 3rd degree heart block).
* History of abnormal life-threatening rhythms as determined by the investigator (e.g., ventricular tachycardia, ventricular fibrillation, 3rd degree heart block)
* Symptomatic (or active) allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis over electrode attachment sites
* Known sensitivity to medical adhesives, isopropyl alcohol, or electrocardiogram (ECG) electrodes including known allergy or sensitivity to fluoroelastomer bands
* Weight more than 180 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Performance in the identification of atrial fibrillation and sinus rhythm | 10 months
  The co-primary endpoints are the sensitivity and specificity in detecting AF from conclusive recordings generated by the software under test, that is recordings resulting in a classification of AF or SR by the SUT, compared to the reference 12-lead ECG.

SECONDARY OUTCOMES:
Evaluation of the classification into heart rate subgroups | 10 months
  The classification into heart rate subgroups will be evaluated for the pairs of strips such that the rhythm classification of the 12-lead ECG is either SR or AF and such that the strip generated by the SUT is classified as either SR or AF and such that the strip generated by the SUT is classified as either SR or AF. The evaluation will be assessed with the concordance of classifications, i.e. the percentage P of identical classifications by the SUT and the reference method, into each of the four following subgroups :
  * SR with a HR between 50 and 99 bpm
  * SR with a HR between 100 and 150 bpm
  * AF with a HR between 50 and 99 bpm
  * AF with a HR between 100 and 150 bpm
Assessment of the clinical equivalence of ECG waveforms | 10 months
  Clinical equivalence of ECG waveforms will be qualitatively and quantitatively assessed between the 6-leads generated by the SUT and the leads I, II, III, aVR, aVL, aVF of the 12-lead ECG by a board of certified cardiologists : The visibility and polarity of the P waves, QRS complexes and T waves will be determined by cardiologists and according to a set of predetermined rules.
Assessment of the clinical equivalence of ECG waveforms | 10 months
  The durations of the QT intervals, QRS complex widths, and PR intervals will be measured by cardiologists with a caliper on the first beat of the 6 marked PQRST complexes and according to a set of predetermined rules for each of the 6 leads of the strips generated by the SUT and the leads I, II, III, aVR, aVL, aVF of the 12-lead ECG.
Determination of the heart rate | 10 months
  The heart rate will be determined by independent cardiologists, or cardiac technicians supervised by cardiologists, from each six-channel strip recorded with the SUT and from each lead I, II, III, aVR, aVL, aVF of the 12-lead strip of the reference ECG. For each simultaneous pair of strips, a reviewer will independently select a common lead with the best signal quality. Then, the reviewer will determine one or several window(s) on the selected lead according to a set of predetermined rules. Finally the number N of complete RR intervals inside these windows and the duration Dt (< 30s) of the windows will be measured with a caliper. The heart rate will then be calculated as 60*N/Dt. The reader-estimated heart rates will later be compared to the heart rates calculated by the SUT

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lellouche, MD, Principal Investigator — Henri Mondor University Hospital
Locations (4):
- Cliniques Universitaires de Bruxelles - Hôpital Erasme, Brussels, Belgium
- France (3):
  - Henri Mondor University Hospital, Créteil, Val De Marne
  - Poitiers University Hospital, Poitiers, Vienne
  - George Pompidou European Hospital, Paris

IPD SHARING:
Plan to Share IPD: No